CLINICAL TRIAL: NCT04133025
Title: Investigation of The Effect of Web-Based System With Oculomotor and Optokinetic Stimulation on Rehabilitation in Vestibular Hypofunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gonulertunc, MSc PT (Specialist Physiotherapist), Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3120598858
Record Dates: First submitted 2019-07-22; First posted 2019-10-21 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Vestibular Rehabilitation; Vestibular Disease
Keywords: Vestibular Rehabilitation; Unilateral vestibular hypofunction
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional vestibular rehabilitation (Active Comparator): Conventional vestibular rehabilitation
  Interventions: Other: Vestibular Rehabilitation
- Vestibular rehabilitation with software (Active Comparator)
  Interventions: Other: Vestibular Rehabilitation

INTERVENTIONS:
Other: Vestibular Rehabilitation — Vestibular Exercises and Software in vestibular rehabilitation

SUMMARY:
The aim of this study was to investigate of the effect of web-based System with oculomotor and optokinetic stimulation on rehabilitation in vestibular hypofunction. In the literature, studies on vestibular rehabilitation in unilateral hypofunction are very limited and there is no study about it.

DETAILED DESCRIPTION:
Vestibular system is one of the sensory systems used for postural control. The function of this system is to maintain balance during head movements and to sense the sense of position in the space.Information from the vestibular system goes to the neural processing center. To achieve or maintain postural control as a result of neural reorganization, balance is achieved by controlling eye movements and muscles.

Basic symptoms in vestibular pathologies are; vertigo and dizziness. Besides these; vestibulo-visual symptoms (oscillopsia, decreased visual acuity, visual tilt, etc.), postural symptoms (feeling of falling, swaying, etc.), and symptoms of motion sickness are. The occurrence of these symptoms varies according to diseases and individual characteristics.

In the treatment of vestibular diseases; there are medical treatment, vestibular rehabilitation, surgical interventions and psychosocial education.Medical treatments; it is often used to suppress or control vestibular symptoms (nausea, etc.). Surgical interventions are the last choice of treatment in patients with severe attacks such as disabling function such as labyrinthectomy or signaling the vestibular nerve. Vestibular Rehabilitation is an exercise based approach to maximize central nervous system compensation for vestibular pathology.

In recent years, the effectiveness of the technologies that have been used in different areas of rehabilitation in vestibular rehabilitation has started to be investigated. In the researches, it is seen that virtual reality is one of the most used technologies. In terms of virtual reality usage, it has cost, size and portability advantages (3). However, in other studies, different systems apart from virtual reality are almost not found among the assistive technologies in vestibular rehabilitation.

In recent years, vestibular rehabilitation methods, adaptation to changing sensory conditions and sensory repetition methods in compensation process have been emphasized to increase adaptation to vestibular losses. However, individual therapeutic programs need to be planned in accordance with clinical symptoms. To this end, there is a need to develop reliable objective and technological feedback techniques to measure the interaction of peripheral senses and central adjustment mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral vestibulopathy between the ages of 18-75,
* No visual disability

Exclusion Criteria:

* Mental retardation,
* Inadequate communication in Turkish;
* Having neurological problems,
* Bilateral vestibular hypofunction
* There is a serious orthopedic problem that will prevent standing and walking.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Change In Results of Head Thrust Test | Eight weeks.
  It tests the vestibulo-ocular reflex (VOR).The examiner holds the patient's head steady in the midline. The patient is instructed to maintain gaze on the nose of the examiner. The examiner then quickly turns the patient's head about 10-15 degrees to one side and observes the ability of the patient to keep the eyes locked on the examiner's nose. the test can also be performed by starting with the head turned to the side, and then making the quick movement back to the midline. If the patient's eyes stay locked on the examiner's nose (i.e., no corrective saccade) , then the peripheral vestibular system is assumed to be intact. Thus in a patient with acute dizziness, the absence of a corrective saccade suggests a Central Neural System(CNS) localization. If, however, the patient's eyes move with the head and then the patient makes a voluntary eye movement back to the examiner's nose (i.e., corrective saccade), then this suggests a lesion of the peripheral vestibular system and not the CNS
Change In Results of Balance Tests At 8 Weeks. | Eight weeks.
  Periodic balance tests are standing on romberg, semi-tandem, tandem, one-leg positions with eyes open and closed in seconds and are recorded by timekeeper.
Change In Levels of Oculomotor Functions | Eight weeks.
  Oculomotor functions are Saccade and Pursuit. They are assessed by software with normal oculomotor frequencies in Hertz.
Change In Results of Head Shake Test at 8 weeks. | Eight weeks.
  The head-shaking test allows determination of an asymmetry between the two horizontal canals [1]. The head of the patient is shaken in the horizontal plane for 20 s and at the end of the stimulation the induced eye movements are observed. If the post head shaking nystagmus is shown, test is positive.
Change In Results of Unterberger Test at 8 weeks | Eight weeks.
  The Unterberger stepping test is a simple means of identifying which labyrinth may be dysfunctional in a peripheral vertigo. The purpose of the Unterberger Test (UT) is to measure asymmetrical vestibulospinal reflex tone resulting from labyrinthine dysfunction. The UT is a low cost evaluation for dizzy patients; however, when compared with gold standard caloric irrigation unilateral weakness (UW) value ≥25%, the UT has not been shown to be a sensitive tool for identifying unilateral vestibular hypofunction

SECONDARY OUTCOMES:
Kinesiophobia Assessment | Before and after eight weeks treatment programmes
  Tampa Kinesiophobia Scale (TKS) is used. It is a 17 item questionnaire used to assess the subjective rating of kinesiophobia or fear of movement. The TSK is a self-completed questionnaire and the range of scores are from 17 to 68 where the higher scores indicate an increasing degree of kinesiophobia.
Quality of Life Assessment: Dizziness Handicap Inventory | Before and after eight weeks treatment programmes
  Dizziness Handicap Inventory is used. The purpose of this scale is to identify difficulties that you may be experiencing because of your dizziness.Item scores are summed. There is a maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional) and a minimum score of 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Physiotherapy and Rehabilitation Doctoral Programme, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Ertunc Gulcelik G, Tarakci D, Gedik Soyuyuce O, Gence Gumus Z, Korkut N, Algun ZC. Research on the Effects of a Web-Based System With Oculomotor and Optokinetic Stimuli on Vestibular Rehabilitation. Am J Phys Med Rehabil. 2021 Jun 1;100(6):555-562. doi: 10.1097/PHM.0000000000001584. PMID 32889859